CLINICAL TRIAL: NCT07027163
Title: Use of Omalizumab in the Treatment of Food Allergy and Anaphylaxis - A Multicenter Retrospective Analysis
Brief Title: A Study About the Use of Omalizumab in the Treatment of Food Allergy and Anaphylaxis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025A2010
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Food Hypersensitivity; Anaphylaxis
Keywords: Food Allergy; IgE-mediated Food Allergy
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Omalizumab Cohort: Adult patients diagnosed with IgE-mediated food allergy who received omalizumab treatment between 2002 and 2022.

SUMMARY:
This was a retrospective, multi-center observational study conducted across four allergy departments in Europe (Berlin, Leipzig, Barcelona, and Basel). The study included patients with immunoglobulin E (IgE)-mediated food allergy who were treated with omalizumab, either as monotherapy or in combination with oral immunotherapy (OIT) between 2002-2022.

ELIGIBILITY:
Inclusion criteria:

* A confirmed history of food allergy, either with or without prior anaphylaxis.
* Treated with omalizumab, either as monotherapy or in combination with OIT.

Exclusion Criteria:

None identified.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients by Response to Treatment | Months 3, 6, 12, and 24
  Patients were classified as treatment responders if an oral food challenge was negative, or a decrease in severity of food allergy during an oral food challenge was determined and no anaphylactic reactions occurred during treatment. Non-responders were those who experienced repetitive food anaphylactic reactions during treatment. Partial treatment responders were patients who experienced less than 1 food anaphylactic reaction despite undergoing treatment.

SECONDARY OUTCOMES:
Frequency of Accidental Reactions | Up to approximately 7 years
  Accidental reactions were those that occurred when a patient unknowingly ingested the food allergen.
Change From Baseline in Allergen Threshold Levels | From Baseline up to approximately 7 years
  Allergen threshold was measured by oral food challenge test. The change in threshold level means the increase in the food dose that the patient was able to tolerate during the food challenge test.
Change From Baseline in Severity of Anaphylactic Reactions | From Baseline up to approximately 7 years
  Change in severity of food allergy was either demonstrated by an oral food challenge or based on the clinical assessment by the investigator.
Health-related Quality of Life (HRQoL) Based on Patient Reported Data as Measured by the EuroQol-5 Dimensions (EQ-5D) Questionnaire | Months 3, 6, 12, and 24
  The EQ-5D is a generic multidimensional measurement tool for describing HRQoL (EuroQol, 1999). The five domains of mobility, self-care ability, daily activities, pain/discomfort and anxiety/depression are considered. For each of the dimensions, the most appropriate answer from three given possibilities is selected (1=no problem, 2=moderate problem, 3=large problem). In addition, the patient marks the current state of health on a scale from 0 (worst conceivable state of health) to 100 (best conceivable state of health). HRQoL was measured if data was available.
HRQoL Based on Patient Reported Data as Measured by the Food Allergy Quality of Life Questionnaire (FAQLQ) | Months 3, 6, 12, and 24
  FAQLQs are disease-specific questionnaires used to measure the impact of food allergy on HRQoL. The forms are completed by the patients themselves or by the parents of food-allergic children and teenagers. Questions are scored on a 7-point scale from 1 (no) to 7 (maximal) impairment on quality of life. HRQoL was measured if data was available.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States